CLINICAL TRIAL: NCT06156969
Title: Muscle Synergies During Gait in Children With Cerebral Palsy Undergoing Robot-assisted Gait Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Paolo Bonato, Director, Motion Analysis Laboratory, Spaulding Rehabilitation Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015P001482
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Results first posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Robotics; Gait rehabilitation
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Robot-assisted gait training (Experimental): Robot-Assisted Gait Training using the LokomatPro device. Total of 18 training sessions, over a period of approximately 6-7 weeks. Sessions will last approximately 60 minutes.
  Interventions: Device: Robot-Assisted Gait Training

INTERVENTIONS:
Device: Robot-Assisted Gait Training — Training will be performed using the LokomatPro. The Lokomat consists of a driven (motorized) gait orthosis (DGO) and an advanced body weight support system, combined with a treadmill. It uses computer-controlled motors which are integrated in the gait orthosis at each hip and knee joint. The exoskeleton is secured to a person's lower limbs using straps.
  Training protocol: Each training session will include 30 minutes of gait training. Training will take over a period of about 6-7 weeks. Sessions will last approximately 60 minutes.

SUMMARY:
This is a single-arm longitudinal study for children with cerebral palsy with gait impairments that involves robot-assisted gait training (RGT) and includes pre and post-data collection visits. The study aims to evaluate changes in muscle synergies in children with Cerebral Palsy (CP) in response to RGT. Additionally, the study aims to investigate the relationship between muscle synergies and the clinical outcomes of RGT.

DETAILED DESCRIPTION:
Participants will be assessed 2 times - before and after training with the robot. All the testing and training sessions will be carried out at Spaulding Rehabilitation Hospital and will include:

Clinical tests:

* A test to evaluate gross motor function
* A test to assess walking speed
* A test to assess endurance

Muscle activity tests:

* A test to derive detailed measures of how well participant walk using a camera-based motion capture system.
* Special sensors (called electromyographic - EMG - sensors) will be used to determine when and how muscles are recruited to generate movements.

Training with the Robot:

Study participants will undergo 18 sessions of robot-assisted gait training for 18 time The training sessions will be carried out by trained study staff. The robot will assist study participants to walk. Each training session will last about 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of spastic cerebral palsy
* 6 to 18 years of age
* Gross Motor Function (GMFCS) Level I, II, III or IV
* Femoral length < size of robotic exoskeleton used for gait training (femur length between 210-350mm)
* Ability to communicate pain or discomfort

Exclusion Criteria:

* Recent use of Lokomat within the last 3 months
* Contraindication to robotic-assisted gait training such us thromboembolic disease, progressive neurologic disorder, cardiovascular or pulmonary contraindications, aggressive behaviors, severe cognitive deficits, bone instabilities, fractures, osteoporosis)
* Skin ulcers in trunk or lower limbs
* Hip, knee, ankle arthrodesis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2018-09-06 (Actual); Study Completion 2020-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Bonato, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Robot-assisted Gait Training: Robot-Assisted Gait Training using the LokomatPro device. Total of 18 training sessions, over a period of approximately 6-7 weeks. Sessions will last approximately 60 minutes.
  Robot-Assisted Gait Training: Training will be performed using the LokomatPro. The Lokomat consists of a driven (motorized) gait orthosis (DGO) and an advanced body weight support system, combined with a treadmill. It uses computer-controlled motors which are integrated in the gait orthosis at each hip and knee joint. The exoskeleton is secured to a person's lower limbs using straps.
  Training protocol: Each training session will include 30 minutes of gait training. Training will take over a period of about 6-7 weeks. Sessions will last approximately 60 minutes.
Period: Overall Study
Arm/Group | Robot-assisted Gait Training
Started | 19
Completed | 13
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.1 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
Gross Motor Function Classification System (GMFCS) [Count of Participants; unit: Participants] — The Gross Motor Function Classification System (GMFCS is a five-level clinical classification system, from the least to the most severe, that describes the gross motor function of children and youth with cerebral palsy based on self-initiated movement abilities and the need for assistive devices such as walkers or wheelchairs. Level I: Walks without limitations; Level II: Walks with limitations; Level III: Walks using a hand-held mobility device; Level IV: Self-mobility with limitations; may use powered mobility; and Level V: Transported in manual wheelchair.
  Participants
    Level I | 2
    Level II | 5
    Level III | 5
    Level IV | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Cosine Similarity of the Muscle Synergies of the Most Affected Lower Limb
Description: Surface electromyographic (EMG) data collected from 16 muscles of the lower limbs during overground gait will be analyzed using the non-negative matrix factorization technique to quantify the patterns of co-activation of muscles. Cosine similarity values will be estimated for the EMG recordings collected pre- and post-intervention. Cosine similarity values will range between 0 and 1, where 1 means that the patterns of co-activation are identical to normative whereas 0 means that they are completely different (as they do not overlap). The percentage of muscle synergies displaying an increase in cosine similarity will be reported.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: Changes in the similarity of muscle synergies recorded from children with CP pre vs post-intervention using normative muscle synergies as a reference
Measure: Mean (Standard Deviation); unit: percentage of muscle synergies
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
percentage of muscle synergies | 2 (6)

2. Secondary Outcome: Change in Gross Motor Function Measure (GMFM) Dimension D
Description: The GMFM Dimension D consists of a battery of thirteen motor tasks that the rater evaluates via visual observation of the motor behavior of the study participant. Dimension D of the scale is focused on standing function. Each item is scored on a 4-point ordinal scale from 0 to 3, where 0 indicates that the participant does not initiate the task; 1 indicates that the participant initiates the task; 2 indicates that the participant partially completes the task; and 3 indicates that the participant completes the task. The minimum value is 0, and the maximum value is 39. Higher values represent better function. The change from baseline to post-intervention is calculated by taking the difference between the value gathered post-intervention and the value gathered pre-intervention.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: Changes in the Gross Motor Function Measure (GMFM) Dimension D score pre- vs post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
units on a scale | 5.9 (8.1)

3. Secondary Outcome: Change in Gross Motor Function Measure (GMFM) Dimension E
Description: The GMFM Dimension E consists of a battery of twenty-four motor tasks that the rater evaluates via visual observation of the motor behavior of the study participant. Dimension E of the scale is focused on walking function. Each item is scored on a 4-point ordinal scale from 0 to 3, where 0 indicates that the participant does not initiate the task; 1 indicates that the participant initiates the task; 2 indicates that the participant partially completes the task; and 3 indicates that the participant completes the task. The minimum value is 0, and the maximum value is 72. Higher values represent a better function. The change from baseline to post-intervention is calculated by taking the difference between the value gathered post-intervention and the value gathered pre-intervention.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: Changes in Gross Motor Function Measure (GMFM) Dimension E pre- vs post-intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
units on a scale | 10.0 (9.3)

4. Secondary Outcome: Percent Change in 10-Meter Walk Test
Description: Study staff will use a stopwatch to measure the time needed by study participants to cover a distance of 10 meters.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: Changes in walking speed relative to baseline (i.e., pre-training)
Measure: Mean (Standard Deviation); unit: percentage of baseline value
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
percentage of baseline value | -0.8 (28.0)

5. Secondary Outcome: Percent Change in 6-Minutes Walk Test
Description: Study staff will measure the distance walked by study participants during an interval of 6 min.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: Changes in endurance as increase in walking distance relative to baseline (i.e., pre-training)
Measure: Mean (Standard Deviation); unit: percentage of baseline walking distance
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
percentage of baseline walking distance | 23.5 (37.7)

6. Secondary Outcome: Percent Change in Edinburgh Visual Gait Scores (EVGS)
Description: The EVGS score is a standardized measure of gait quality derived using criteria based on visual observation of gait patterns in children with cerebral palsy. The EVGS includes 17 gait parameters and uses a three-point ordinal scale for each parameter, corresponding to normal, moderate, and severe deviation, respectively. The total score range is from 0 to 34 points, where 0 corresponds to normal gait and greater than 0 indicates gait abnormality.
Time Frame: Data collected at baseline and at completion of the 7-week intervention
Population: Changes in quality of gait as captured by the Edinburgh Visual Gait Scores (EVGS) relative to baseline (i.e., pre-training) value
Measure: Mean (Standard Deviation); unit: percentage of baseline value
Arm/Group | Robot-assisted Gait Training
Number analyzed (Participants) | 13
percentage of baseline value | 16.7 (12.7)

ADVERSE EVENTS:
Time Frame: From baseline to study completion, on average 7 weeks.
Arm/Group | Robot-assisted Gait Training
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT06156969/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/69/NCT06156969/SAP_001.pdf